CLINICAL TRIAL: NCT01042054
Title: The Effects of Local Infiltration Versus Epidural on Recovery
Brief Title: Comparison of Analgesic Methods, and Their Effects on Patient Recovery, Following Liver Surgery
Acronym: LIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Erica Revie, Miss Erica Revie, University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09/S1102/17; 2009/R/SU/04 (Other: South East Scotland Research Ethics Committee 02)
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Postoperative Pain
Keywords: Postoperative Care; Enhanced; Recovery; Hepatectomy; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural (Active Comparator): Patients will follow a standard optimised recovery protocol, including epidural analgesia for the first 48 hours postoperatively.
  Interventions: Other: Standard optimised recovery protocol.
- Wound catheter (Experimental): Patients will follow a standard optimised recovery protocol, but analgesia in the first 48 hours will be delivered through local anaesthetic wound catheters and additional patient-controlled analgesia, instead of epidural analgesia.
  Interventions: Other: Wound catheter plus patient-controlled analgesia.

INTERVENTIONS:
Other: Standard optimised recovery protocol. — * Epidural analgesia for the first 48 hours postoperatively.
  * Sham wound catheter attached to anterior abdominal wall, for purposes of blinding.
  * Standard oral analgesic regime commenced at 48 hours, and continued until discharge from hospital.
  * Optimised recovery protocol followed throughout.
  Arms: Epidural
Other: Wound catheter plus patient-controlled analgesia. — * Continuous infusion of local anaesthetic administered via wound catheters for the first 48 hours postoperatively.
  * Additional patient-controlled intravenous opiate analgesia available to patient during this time period.
  * Sham epidural catheter applied to the patient's back for purposes of blinding.
  * Standard oral analgesic regime commenced at 48 hours, and continued until discharge from hospital.
  * Optimised recovery protocol followed throughout.
  Other Names: ON-Q PainBuster
  Arms: Wound catheter

SUMMARY:
The provision of adequate pain relief following major liver surgery is essential, not only for patient comfort, but for the prevention of complications, such as chest infection.

Commonly, pain relief in the first few days after surgery is provided by epidural analgesia. Drugs are delivered to the area around the spinal cord, through a fine plastic tube placed in the patients back, and this blocks sensation from the abdomen downwards, thereby providing effective pain relief without the need for opiate analgesia (e.g. morphine). Opiate analgesia can cause nausea, drowsiness and constipation, and its use should be minimised. Epidurals, however, can be associated with some problematic side effects. Low blood pressure is commonly encountered, and not only can its treatment be associated with complications, but patients are often confined to bed.

Mobility can also be limited if muscle function in the legs, (in addition to sensation), is inadvertently affected by the epidural drugs. Other problems associated with epidural use are the relatively common failure of the technique to provide adequate analgesia (20%), and some extremely rare but potentially disastrous complications of epidural insertion.

An alternative technique, is the provision of pain relief directly into the wound, via one or more multi-holed tubes(catheters), placed either in or close to the wound. This technique alone does not provide as effective analgesia as a functioning epidural, but when combined with other intravenous or oral analgesia, has been shown to be effective following a variety of surgical procedures.

It is hypothesised that, following major liver surgery, the use of this latter technique may result in superior outcome and faster recovery, when compared with epidural, by avoidance of the side effects and complications discussed above.

In this study, patients scheduled to undergo major liver surgery at the Royal Infirmary of Edinburgh with be randomly assigned to receive the first two days of pain relief either by epidural, or by wound catheter plus additional analgesia. Both groups will then receive an identical oral analgesic regime for the remainder of the hospital stay.

Outcomes of interest will include the quality of pain relief attained, patient mobility, frequency of complications, and overall recovery time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open hepatic resection for benign or malignant conditions.
* Able to understand the nature of the study and what will be required of them.
* Men and non-pregnant, non-lactating women.
* BMI 18-40.

Exclusion Criteria:

* Patients with contraindication to either epidural or wound catheter techniques.
* Inability to give written, informed consent.
* Patients with dementia or neurological impairment.
* Patients with pre-existing condition limiting mobility.
* Underlying cirrhotic liver disease.
* Jaundice (Bilirubin > 50 μmol/L).
* Liver resection combined with secondary surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Length of time to reach criteria for discharge from hospital. | This will be assessed twice daily until criteria for dicharge from hospital are met.

SECONDARY OUTCOMES:
Pain scores, assessed using numerical rating score (0 to 10). | Assessed at 2, 6 & 12 hours following closure of wound, and daily thereafter until discharge from hospital, or day 7, whichever is sooner.
Nausea and sedation scores, assessed using numerical rating score (0 to 3). | Assessed at 2, 6 & 12 hours following closure of wound, and daily thereafter until discharge from hospital, or day 7, whicever is sooner.
Sleep disturbance, assessed using numerical rating score (0 to 10). | Assessed daily from the morning following surgery until discharge from hospital, or day 7, whichever is sooner.
Volume of intravenous fluids received in the first 48 hours following operation (ml). | Data collected daily for first 48 hours following operation.
Mobility (percentage of time spent lying / sitting, standing or walking, as measured by ActivPAL meter). | From the end of the operative procedure until discharge from hospital, or day 7, whichever is sooner.
Time to return of bowel function (days). | Assessed daily until return of bowel function.
Length of time to meet criteria for discharge from the High Dependency Unit. | Assessed twice daily until criteria for discharge from the High Dependency Unit met.
Complications (General and Technical). | Assessed daily throughout hospital admission, and at outpatient review clinic 4-6 weeks following discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Erica J Revie, Principal Investigator — University of Edinburgh
Locations (1):
- Department of Surgery, Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Derived] Revie EJ, McKeown DW, Wilson JA, Garden OJ, Wigmore SJ. Randomized clinical trial of local infiltration plus patient-controlled opiate analgesia vs. epidural analgesia following liver resection surgery. HPB (Oxford). 2012 Sep;14(9):611-8. doi: 10.1111/j.1477-2574.2012.00490.x. Epub 2012 Jun 10. PMID 22882198